CLINICAL TRIAL: NCT04891471
Title: WHOle Brain Irradiation and STEreotactic Radiosurgery for Five or More Brain Metastases (WHOBI-STER): a Prospective Comparative Study of Neurocognitive Outcomes, Level of Autonomy in Daily Activities and Quality of Life
Brief Title: WHOle Brain Irradiation or STEreotactic Radiosurgery for Five or More Brain Metastases (WHOBI-STER)
Acronym: WHOBI-STER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mediterranean Institute of Oncology (Other)
Collaborators: University of Messina (Other); University of Palermo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70/2020/CECT2
Record Dates: First submitted 2021-04-20; First posted 2021-05-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Neurocognitive Deficit; Quality of Life; Activities of Daily Living
Keywords: multiple brain metastasis; neurocognitive decay; whole brain radiotherapy; stereotactic radiosurgery; stereotactic body radiotherapy; quality of life; solid tumor; Activities of Daily Living; best supportive care; palliative radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRS/SBRT arm (Experimental): Patients with five or more brain metastasis assigned by randomization to Stereotactic RadioSurgery (SRS) or Stereotactic Body RadioTherapy (SBRT) will be treated with a highly-conformal metastasis-directed single dose between 15 and 24 Gy or fractionated dose (e.g. 27 Gy in 3 fractions), respectively, depending on lesion size, while sparing clinically negative brain. The treatment will be delivered using five non-coplanar arcs and a mono-isocentric technique.
  Interventions: Radiation: Stereotactic RadioTherapy
- WBI arm (Active Comparator): Patients with five or more brain metastasis assigned by randomization to Whole Brain Irradiation (WBI) will be treated using a 3D-Conformal RadioTherapy technique for a uniform dose delivery of 30 Gy in 10 daily/fractions to the target, that is entire brain.
  Interventions: Radiation: Whole Brain Irradiation

INTERVENTIONS:
Radiation: Stereotactic RadioTherapy — To treat only brain metastasis identified through Magnetic Resonance imaging by means of stereotactic radiotherapy (experimental intervention) to determine if sparing of clinically uninvolved brain implies a better neurocognitive performance, quality of life and level of autonomy in activities of daily living respect to Whole Brain Irradiation (active comparator).
  Other Names: Stereotactic RadioSurgery; Stereotactic Body RadioTherapy
  Arms: SRS/SBRT arm
Radiation: Whole Brain Irradiation — To irradiate the entire brain, site of at least 5 parenchymal metastasis.
  Other Names: Whole Brain Radiotherapy, Panencephalic Radiotherapy
  Arms: WBI arm

SUMMARY:
This work aims to evaluate neurocognitive performance, daily activity and quality of life and local control among patients with brain metastasis (MBM) ≥ 5 due to solid tumors treated with Stereotactic RadioSurgery (SRS) or Whole Brain RadioTherapy (WBRT). This multicentric randomised controlled trial will be conducted at the Fondazione IOM (Viagrande) in collaboration with REM (Viagrande), Hospital G. Martino (Messina) and Hospital Civico ARNAS (Palermo). It will involve, within 5 years starting from 15 September 2020, the enrollment of 100 patients (50 for each arm) with MBM ≥ 5, age ≥ 18 years, Karnofsky Performance Status (KPS) ≥ 70, life expectancy > 3 months, histological confirmation of primary tumor, with controlled or controllable extracranial disease, baseline Montreal Cognitive Assessment (MoCA) of 20/30, Barthel Activities of Daily Living score 90/100, to be subjected to SRS on each brain lesion by LINAC with monoisocentric technique and non-coplanar arcs (experimental arm) or to WBRT (control arm). The primary endpoints are neurocognitive performance, quality of life and autonomy in daily-life activities variations, the first one assessed by Moca Score and Hopkins Verbal Learning Test - Revised, the second one through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 Palliative Care (EORTC QLQ-C15-PAL) and Brain Neoplasm (BN-20) questionnaires, the third one through the Barthel Index, respectively. The secondary endpoints are time to intracranial failure, overall survival, retreatments frequency, acute and late toxicities, KPS decrease. It will be considered significant a statistical difference of at least 29% between the two arms (statistical power of 80% with a significance level of 95%). This trial has been approved by the local ethics committee on July 7th 2020 (record 70). Several studies debate what is the predominant factor accountable for the development of neurocognitive decay among patients undergoing brain irradiation for MBM: radiotherapy, especially if extended to the entire brain, or intracranial disease progression? Answer to this question may come from current opportunity, thanks to recent technological advancement, to treat, with significant time savings, improved patient comfort and at the same time minimizing the dose to healthy brain tissue, Multiple Brain Metastasis simultaneously, otherwise attackable only by panencephalic irradiation. The pursuit of a local control rate comparable to that obtainable with WBRT remains the fundamental prerequisite for the aforementioned related assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Life expectancy > 3 months
* Brain metastases number ≥ 5
* Primary tumor histologic diagnosis
* Complete Extracranial staging
* Montreal Cognitive Assessment ≥ 20/30
* Barthel Activities of Daily Living ≥ 90/100
* KPS ≥ 70
* Signed Informed Consent

Exclusion Criteria:

* Brain-MRI contraindications
* Contraindications to SRS
* Pregnancy
* Hemorrhagic cerebral disease
* Miliary metastases
* Massive perilesional edema
* Leptomeningeal involvement
* Previous brain irradiation
* Dementia
* Non-solid brain tumor
* Ischaemic event
* Alcohol and/or drugs abuse
* Anxiety and depression
* KPS ≤ 60
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive changes detected through Moca Score | Change from Baseline pre-Radiotherapy Neurocognitive Functional Status every three months after treatment through study completion, an average of 1 year
  To assess how neurocognitive performance changes after SRS/SBRT compared to WBI
Changes of Autonomy in daily activities detected through the Barthel Index | Change from Baseline pre-Radiotherapy Barthel Index every three months after treatment through study completion, an average of 1 year
  To assess how level of autonomy in activities of daily living changes after SRS/SBRT compared to WBI
Change in quality of life detected though the EORTC QLQ-C15-PAL questionnaire | Change from Baseline pre-Radiotherapy EORTC QLQ-C15-PAL questionnaire every three months after treatment through study completion, an average of 1 year
  To assess how quality of life changes after SRS/SBRT compared to WBI
Neurocognitive changes detected through Hopkins Verbal Learning Test - Revised | Change from Baseline pre-Radiotherapy Neurocognitive Functional Status every three months after treatment through study completion, an average of 1 year
  To assess how neurocognitive performance changes after SRS/SBRT compared to WBI
Change in quality of life detected though the BN-20 questionnaire | Change from Baseline pre-Radiotherapy BN-20 questionnaire every three months after treatment through study completion, an average of 1 year
  To assess how quality of life changes after SRS/SBRT compared to WBI

SECONDARY OUTCOMES:
Time to local failure | every three months after treatment through study completion, an average of 1 year
  Time between treatment and cerebral disease progression detected through Magnetic Resonance imaging
Overall Survival | after treatment completion through study completion, an average of 1 year
  Time from the first day of treatment to exitus
Re-treatment rate | after first treatment completion through study completion, an average of 1 year
  Difference in needing further subsequent radiotherapy treatment between SRS/SBRT and WBI arms
Acute Central Nervous System (CNS) toxicities evaluated by means of Radiation Therapy Oncology Group (RTOG)/ European Organization for Research and Treatment of Cancer (EORTC) Radiation Toxicity Grading | from treatment completion until three months later
  Toxicities registered within three months from treatment
Late Central Nervous System (CNS) toxicities evaluated by means of Radiation Therapy Oncology Group (RTOG)/ European Organization for Research and Treatment of Cancer (EORTC) Radiation Toxicity Grading | from three months after treatment completion through study completion, an average of 1 year
  Toxicities registered after three months from treatment
Karnofsky Performance Status changing | after treatment completion through study completion, an average of 1 year
  Evaluation of how patient's performance status modifies after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ferini, Principal Investigator — REM Radiotherapy (parent company of Mediterranean Institute of Oncology)
Locations (4):
- Italy (4):
  - Fondazione Istituto Oncologico del Mediterraneo, Viagrande, Catania
  - REM Radiotherapy (parent company of Mediterranean Institute of Oncology), Viagrande, Catania
  - Radiation Oncology Unit - Department of Biomedical, Dental Science and Morphological and Functional Images, University of Messina, Messina
  - Radiation Oncology, ARNAS-Civico Hospital, Palermo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Ferini G, Viola A, Valenti V, Tripoli A, Molino L, Marchese VA, Illari SI, Rita Borzi G, Prestifilippo A, Umana GE, Martorana E, Mortellaro G, Ferrera G, Cacciola A, Lillo S, Pontoriero A, Pergolizzi S, Parisi S. Whole Brain Irradiation or Stereotactic RadioSurgery for five or more brain metastases (WHOBI-STER): A prospective comparative study of neurocognitive outcomes, level of autonomy in daily activities and quality of life. Clin Transl Radiat Oncol. 2021 Dec 2;32:52-58. doi: 10.1016/j.ctro.2021.11.008. eCollection 2022 Jan. PMID 34926839